CLINICAL TRIAL: NCT04572672
Title: Effect of Pursed-Lip Breathing Combined With Number Counting on Blood Pressure and Heart Rate in Hypertensive Urgency Patients: A Randomized Controlled Trial
Brief Title: Effect of Pursed-Lip Breathing on Blood Pressure and Heart Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Praew Kotruchin, Assistant professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HE611586
Record Dates: First submitted 2020-09-17; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Hypertensive Urgency
Keywords: Hypertensive crisis; Uncontrolled hypertension; Mindfulness; Slow breathing; Emergency room
MeSH Terms: conditions — Hypertensive Crisis; Hypoventilation; Emergencies

STUDY DESIGN:
Intervention Model Description: This was a single-blinded randomized controlled trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Purse lip breathing with number counting arm (Active Comparator): 1) Position: The patient lies down in a semi-supine position, the bed is adjusted by 45-60 degrees, 2) Pursed-lip breathing and number counting "one and two" during inspiration, and 3) Number counting, "one, two, three, and four" during exhalation for the first 15 minutes (min) of each hour, total study time was 3 hours or until the patient was discharged from the ER.
  Interventions: Other: Non-pharmacologic treatment; Pursed-Lip Breathing Combined with Number Counting
- Control arm (No Intervention): The patients who were allocated to the control group received usual nursing care i.e. bed rest in a supine position in a quiet area. Patients were advised to limit their activity. The frequency of the vital signs monitoring and pharmacologic treatment were the same as the intervention group.

INTERVENTIONS:
Other: Non-pharmacologic treatment; Pursed-Lip Breathing Combined with Number Counting — Pursed-lip breathing and number counting "one and two" during inspiration, and then number counting, "one, two, three, and four" during exhalation. The nurse advised the patient to continue pursed-lip breathing with number counting for the first 15 minutes (min) of each hour to prevent the patient from being exhausted, total study time was 3 hours, or until the patient was discharged from the ER, or was withdrawn from the study.
  Arms: Purse lip breathing with number counting arm

SUMMARY:
Hypertensive urgency (HT urgency) is an alarm sign of uncontrolled hypertension. It can be aggravated by nonadherent to medication and psychosocial stress. Mindfulness is beneficial for reducing stress, while deep and slow breathing is effective for blood pressure (BP) lowering. The objective of the study was to assess the effect of pursed-lip breathing with number counting (PLB with NC) that promotes mindfulness and a deep/slow breathing pattern on BP and heart rate (HR) in the HT urgency patients.

DETAILED DESCRIPTION:
This was a single-blinded randomized controlled trial. Patients aged between 18-80 years old, diagnosed with HT urgency, who presented at the emergency room of Srinagarind hospital (a 1000-bed, tertiary-care level university hospital), Khon Kaen University between September 1st, 2019 to June 30th, 2020, were enrolled. Those with cardiac arrhythmias, acute HF, acute coronary syndromes, acute stroke, acute respiratory failure, alteration of consciousness, and pregnant women were excluded. This study was approved by the Khon Kaen University Ethical Review Board in Human Research (HE611586). All patients gave their written informed consent before the enrollment.HT urgency was defined as SBP >180 mmHg and/or DBP >110 mmHg without any signs or symptoms of target organ damages.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old patients who diagnosed with HT urgency, who presented at the emergency room

Exclusion Criteria:

* Patients with cardiac arrhythmias,
* Acute heart failure
* Acute coronary syndromes
* Acute stroke
* Acute respiratory failure
* Alteration of consciousness
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Change of systolic blood pressure | pre-intervention and 3 hours after the intervention
  The change of systolic blood pressure level was assessed.
Change of diastolic blood pressure | pre-intervention and 3 hours after the intervention
  The change of diastolic blood pressure level was assessed.
Change of heart rate | pre-intervention and 3 hours after the intervention
  The change of heart rate was assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Khon Kaen Unversity, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No